CLINICAL TRIAL: NCT06841640
Title: Two-part, Single-dose, Dose-finding Study to Assess the Safety, Tolerability, Pharmacokinetics and Bronchodilator Effects of AERO-007 Inhalation Solution Using a General Purpose Nebulizer in Healthy Volunteers and Subjects With COPD
Brief Title: Phase 1/Phase 2a Study of AERO-007 Inhalation Solution, a Nebulized LABA/LAMA Combination for Maintenance Treatment of COPD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AeroRx Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: AERO-007-01
Record Dates: First submitted 2025-02-14; First posted 2025-02-24 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: COPD
Keywords: LABA; LAMA; LABA/LAMA; Inhalation; Nebulization; COPD; HVs; Single-dose; Crossover; Randomized; Placebo-controlled; Bronchodilation; FEV1; Indacaterol; Glycopyrrolate
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Two cohort study. Cohort 1 is open-label, four-way crossover in 8 healthy subjects; Cohort 2 is double-blind, three-way crossover in 16 COPD patients.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- AERO-001 low dose (Experimental)
  Interventions: Drug: AERO-001
- AERO-001 high dose (Experimental)
  Interventions: Drug: AERO-001
- AERO-002 low dose (Experimental)
  Interventions: Drug: AERO-002
- AERO-002 high dose (Experimental)
  Interventions: Drug: AERO-002
- AERO-007 low dose (Experimental)
  Interventions: Drug: AERO-007
- AERO-007 high dose (Experimental)
  Interventions: Drug: AERO-007
- Placebo (Experimental)
  Interventions: Drug: AERO-007

INTERVENTIONS:
Drug: AERO-001 — Open-label
  Other Names: Part 1
  Arms: AERO-001 high dose; AERO-001 low dose
Drug: AERO-002 — Open-label
  Other Names: Part 1
  Arms: AERO-002 high dose; AERO-002 low dose
Drug: AERO-007 — Double-blind
  Other Names: Part 2
  Arms: AERO-007 high dose; AERO-007 low dose; Placebo

SUMMARY:
This is a phase 1/phase 2a, single dose, crossover study conducted in two parts.

Part 1: Phase 1, open-label, 4-period crossover study in 8 healthy subjects to determine the optimal dose of AERO-001 and AERO-002, the active components of AERO-007 combo bronchodilator, using the systemic pharmacokinetic (PK) profile.

Part 2: Phase 2a, randomized, double-blind, placebo-controlled, 3-period crossover study in 16 subjects with COPD to determine the safety, tolerability, PK, and bronchodilator profile of AERO-007 inhalation solution administered via oral inhalation using a general-purpose nebulizer.

DETAILED DESCRIPTION:
According to the Global Initiative for Chronic Obstructive Lung Disease [GOLD] guidelines, combination of a long-acting beta-agonist (LABA) bronchodilator and a long-acting muscarinic antagonist (LAMA) bronchodilator is the preferred choice for initial pharmacotherapy for COPD patients with high symptom severity, frequently experiencing breathlessness and patients with high exacerbation risk.

Although there are currently multiple LABA+LAMA combination bronchodilators available in an inhaler (MDI, DPI, and SMI), a significant number of COPD patients, generally high risk and older patients, do not receive optimal benefit from inhalers. Nebulized delivery provides an effective alternative for these patients. Currently there are no approved LABA+LAMA combinations available for nebulization delivery.

AERO-007 is a propriety inhalation solution formulation of fixed-dose combination of LABA+LAMA (indacaterol, AERO-001 and glycopyrrolate, AERO-002) under development for delivery using a general purpose nebulizer.

This study consists of two parts. In Part 1 (Phase 1), 8 healthy subjects will be randomized to receive single doses of 4 study treatments in an open-label, crossover design (low and high doses of AERO-001 and AERO-002). In Part 2 (Phase 2a), 16 subjects with clinically stable COPD will be randomized to receive single doses of 3 study treatments in a double-blind, crossover design (low and high doses of AERO-007 and placebo) administered by random sequence.

ELIGIBILITY:
Cohort 1 (Healthy Subjects)

Inclusion Criteria:

* Male or female aged 18 to 55 years
* FEV1 > 80% of predicted normal (using the Global Lung Function Initiative GLI 2012 reference values)
* Body mass index > 18 and < 32 kg/m2
* Female subjects of childbearing potential must not be pregnant, breast feeding or lactating and use, with their partner, a male condom plus an approved method of highly effective birth control method
* Female subjects of childbearing potential must have a negative serum or urine pregnancy test at the Screening Visit
* Male subjects who are sexually active with a partner of childbearing potential must use, with their partner, a male condom plus an approved method of highly effective contraception from the time of informed consent
* Participants must be in good health as determined by medical history, physical examination, vital signs, 12-lead ECG and clinical laboratory assessments at the time of screening, as judged by the Investigator
* Willing and able to provide written informed consent

Exclusion Criteria:

* Any condition or abnormality (including medical history, clinical laboratory, ECG, physical examination, or vital sign abnormalities), current or past, that, in the opinion of the Investigator
* Lower respiratory tract infection within 6 weeks prior to the Screening Visit
* History of malignancy of any organ system, except for localized skin cancers, within 5 years prior to the Screening Visit
* Major surgery (requiring general anaesthesia) within 6 weeks prior to the Screening Visit
* Positive serum hepatitis B surface antigen (HbsAg), hepatitis C virus antibodies (HCV Ab) or human immunodeficiency virus (HIV) 1 and/or 2 antibodies
* Chronic viral infection or immunodeficiency condition
* History of any drug and/or alcohol abuse in the past 2 years
* Current or previous use of tobacco, nicotine products or e-cigarettes within 6 months
* Smoking history of > 5 pack years
* Regular alcohol consumption in males >21 units per week and females >14 units per week
* Positive urine drugs of abuse test and/or alcohol breath test
* Donation of 450 mL of blood within 8 weeks
* Known hypersensitivity to any ingredients in the formulation for AERO-001, AERO-002, and AERO-007
* Participation in another investigational drug study within 30 days, 5 half-lives or twice the duration of the biological effect

Cohort 2 (Subjects with COPD)

Inclusion Criteria:

* Male or female aged 40 to 75 years
* Clinical diagnosis of COPD according to the Global Initiative for Chronic Obstructive Lung Disease [GOLD] Report, 2024 for at least 12 months
* Post-bronchodilator spirometry (within 30 minutes following 4 puffs of salbutamol) demonstrating the following:
* FEV1 > 40 and < 80% of predicted normal (using the Global Lung Function Initiative GLI 2012 reference values)
* FEV1/FVC ratio < 0.70
* ≥ 150 mL increase from pre-bronchodilator FEV1
* Ability to change current COPD therapy and discontinue long-acting bronchodilators for the duration of the study and short-acting bronchodilators for 8 hours prior to dosing at each treatment visit
* Current or former-smokers with at least 10 pack-year smoking history (eg, at least 1 pack/day for 10 years, 10 packs/day for 1 year)
* Ability to perform reproducible spirometry according to the American Thoracic Society (ATS)/European Respiratory Society (ERS) guidelines
* Female subjects of childbearing potential must not be pregnant, breast feeding or lactating and use, with their partner, a male condom plus an approved method of highly effective birth control method
* Willing and able to provide written informed consent

Exclusion Criteria:

* Female subjects who are pregnant, breast-feeding or lactating
* Current evidence or recent history of significant comorbidities; including cardiovascular disease (such as myocardial infarction, cardiac failure, uncontrolled hypertension, or life-threatening arrhythmias), uncontrolled diabetes, neurologic, psychiatric, hepatic, renal, immunological, or haematological conditions within the last 6 months
* Positive serum HbsAg, HCV Ab or HIV 1 and/or 2 antibodies
* Lower respiratory tract infection within 6 weeks
* Recent history of hospitalization due to an exacerbation of airway disease or acute worsening of COPD requiring antibiotic or corticosteroid treatment within 6 months
* Other respiratory disorders: Current diagnosis of predominant asthma, lung cancer, bronchiectasis, interstitial lung disease, tuberculosis, pulmonary hypertension, or other non-specific pulmonary diseases
* Prior lung volume reduction surgery or history of chest/lung irradiation
* Daily oxygen therapy for > 12 hours per day
* Body mass index >35 kg/m2
* Current or recent history of medical conditions that are contraindicated for use of an inhaled LAMA (such as urinary retention or bladder neck obstruction type symptoms, prostatic hypertrophy, or narrow-angle glaucoma) within the last 6 months
* Current or recent history (previous 12 months) of excessive use or abuse of alcohol (males >21 units per week and females >14 units per week)
* Current evidence or history (within the past 2 years) of abusing legal drugs or use of illegal drugs or substances
* Donation of 450 mL of blood within 8 weeks
* Major surgery (requiring general anaesthesia) within 6 weeks
* History of malignancy of any organ system, except for localized skin cancers, within 5 years
* Known hypersensitivity to any ingredients in the formulation for AERO-001, AERO-002, and AERO-007
* Participation in another investigational drug study within 30 days, 5 half-lives or twice the duration of the biological effect, whichever is longer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-06-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - AUC | Day 1
  AUC0-t (Area under the plasma concentration from time 0 to the last collection time)
Pharmacokinetics - Cmax | Day 1
  Cmax (Maximum plasma concentration)
Bronchodilation - FEV1 | Day 1
  Change from baseline in actual FEV1 over 12 hours
Bronchodilation - FEV1 AUC | Day 1
  FEV1 AUC (0-12 hours)
Bronchodilation - Peak FEV1 | Day 1
  Peak FEV1 (0-4 hours)

SECONDARY OUTCOMES:
Adverse events | From the first dose to the end of study
  Treatment-emergent AEs

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, MD, Principal Investigator — Medicines Evaluation Unit Ltd
Locations (1):
- Medicines Evaluation Unit Ltd, Manchester, United Kingdom